CLINICAL TRIAL: NCT00612261
Title: Arteriovenous Crossing Sheathotomy Versus Intravitreal Triamcinolone Acetonide Injection for Treatment of Macular Edema Associated With Branch Retinal Vein Occlusion
Brief Title: Sheathotomy vs. Intravitreal Triamcinolone for Branch Retinal Vein Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Hyoung Jun Koh, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: koh003
Record Dates: First submitted 2008-01-25; First posted 2008-02-11 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-01

CONDITIONS: Macular Edema; Branch Retinal Vein Occlusion
Keywords: Branch retinal vein occlusion; treatment
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The group 1 patients receive AV sheathotomy for macular edema secondary to branch retinal vein occlusion.
  Interventions: Procedure: Arteriovenous Crossing Sheathotomy
- 2 (Active Comparator): The group 2 patients receive IVTA.
  Interventions: Procedure: Intravitreal Triamcinolone Acetonide Injection

INTERVENTIONS:
Procedure: Arteriovenous Crossing Sheathotomy — In each sheathotomy patient, a standard pars plana vitrectomy is performed, followed by surgical separation of the posterior cortical vitreous from the optic nerve and posterior retina. After the relevant arteriovenous crossing site is identified based on preoperative FA, a bent microvitreoretinal blade is used to open the internal limiting membrane and the nerve fiber layer over the artery, with the incision commencing 100-200 micrometer proximal to the AV crossing. The incision is continued parallel to and under the retinal arteriole, with a gentle lifting motion, until the common AV crossing sheath is encountered and incised in a side-to-side manner. The completion of AV dissection is confirmed by an elevation of the overlying artery.
  Arms: 1
Procedure: Intravitreal Triamcinolone Acetonide Injection — The IVTA group receive intravitreal injection of 4 mg/0.1 mL triamcinolone acetonide (40 mg/mL; Tamceton®; Hanall Pharmaceutical, Seoul, Korea). The injections are performed using 0.5% proparacaine drops (Alcaine®; Alcon Laboratories, Fort Worth, TX) for topical anesthesia under sterile conditions. The drug is injected through the inferotemporal pars plana using a 30-gauge needle. The correct intravitreal localization of the suspension, and perfusion of the optic nerve head, are then confirmed by indirect ophthalmoscopy.
  Arms: 2

SUMMARY:
Branch retinal vein occlusion (BRVO) is a common retinal vascular disease occurring in a significant number of individuals older than 50 years.The most common cause of visual disturbance in BRVO patients is macular edema, which has been reported in 60% of patients. Macular grid laser photocoagulation has been shown to be effective in the treatment of macular edema arising from BRVO. Some eyes are resistant to conventional grid laser treatment, and the conventional treatment is not useful in patients with intraretinal hemorrhages that may interfere with laser photocoagulation. Moreover, several studies have shown that conventional grid laser treatment for macular edema may be associated with complications.

Intravitreal triamcinolone acetonide (IVTA) injection has recently been reported to be effective in the treatment of macular edema of various etiologies.On the other hand, arteriovenous sheathotomy is a surgical method suggested for treatment of macular edema in BRVO patients, and has been reported to be efficacious in patients refractory to conventional focal or grid laser macular photocoagulation.Both treatment modalities have been reported to be associated with reductions in central macular thicknesses and improved visual acuities.

The purpose of the study is to compare the efficacies of arteriovenous (AV) sheathotomy and intravitreal triamcinolone (IVTA) injection in the treatment of macular edema associated with branch retinal vein occlusion (BRVO).

ELIGIBILITY:
Inclusion Criteria:

* recent onset (within the 6 months prior to enrollment) of macular edema resulting from BRVO
* best corrected Early Treatment Diabetic Retinopathy Study (ETDRS) scores ≤ 40 letters (Snellen equivalent ≤ 20/40
* intraretinal hemorrhages involving the foveal centers
* generalized breakdown of the inner blood-retina barrier, as documented by diffuse fluorescein leakage on angiography, or diffuse thickening of the retina on optical coherence tomography (OCT), with involvement of the foveal center and most of the macular area, and with foveal thicknesses ≥ 250 micrometer

Exclusion Criteria:

* prior history of intraocular surgery including cataract extraction
* prior history of laser treatments including panretinal photocoagulation and focal/grid macular photocoagulation
* prior history of elevated intraocular pressure secondary to steroid treatment
* prior history of glaucoma or ocular hypertension
* presence of comorbid ocular conditions that might affect visual acuity (VA).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
best-corrected ETDRS visual acuity score | baseline, at 1,3,6 months after either treatment

SECONDARY OUTCOMES:
complication rate | at 1,3,6 months after either treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jun Koh, MD, PhD, Principal Investigator — Yonsei University Heath System
Locations (1):
- Yonsei University Health System, Seoul, South Korea

REFERENCES:
- [Background] Parodi MB, Spasse S, Iacono P, Di Stefano G, Canziani T, Ravalico G. Subthreshold grid laser treatment of macular edema secondary to branch retinal vein occlusion with micropulse infrared (810 nanometer) diode laser. Ophthalmology. 2006 Dec;113(12):2237-42. doi: 10.1016/j.ophtha.2006.05.056. Epub 2006 Sep 25. PMID 16996596
- [Background] Chen SD, Sundaram V, Lochhead J, Patel CK. Intravitreal triamcinolone for the treatment of ischemic macular edema associated with branch retinal vein occlusion. Am J Ophthalmol. 2006 May;141(5):876-883. doi: 10.1016/j.ajo.2005.12.011. Epub 2006 Mar 9. PMID 16527226
- [Background] Lee H, Shah GK. Intravitreal triamcinolone as primary treatment of cystoid macular edema secondary to branch retinal vein occlusion. Retina. 2005 Jul-Aug;25(5):551-5. doi: 10.1097/00006982-200507000-00001. PMID 16077348
- [Background] Chalam KV, Shah GY, Shah VA. Vitrectomy with or without arteriovenous adventitial sheathotomy for macular edema associated with branch retinal vein occlusion. Am J Ophthalmol. 2005 Jun;139(6):1146; author reply 1146-7. doi: 10.1016/j.ajo.2005.02.024. No abstract available. PMID 15953467
- [Background] Hayashi K, Hayashi H. Intravitreal versus retrobulbar injections of triamcinolone for macular edema associated with branch retinal vein occlusion. Am J Ophthalmol. 2005 Jun;139(6):972-82. doi: 10.1016/j.ajo.2004.12.087. PMID 15953425
- [Background] Horio N, Horiguchi M. Effect of arteriovenous sheathotomy on retinal blood flow and macular edema in patients with branch retinal vein occlusion. Am J Ophthalmol. 2005 Apr;139(4):739-40. doi: 10.1016/j.ajo.2004.10.026. PMID 15808186
- [Background] Lakhanpal RR, Javaheri M, Ruiz-Garcia H, De Juan E Jr, Humayun MS. Transvitreal limited arteriovenous-crossing manipulation without vitrectomy for complicated branch retinal vein occlusion using 25-gauge instrumentation. Retina. 2005 Apr-May;25(3):272-80. doi: 10.1097/00006982-200504000-00004. PMID 15805902
- [Background] Ozkiris A, Evereklioglu C, Erkilic K, Ilhan O. The efficacy of intravitreal triamcinolone acetonide on macular edema in branch retinal vein occlusion. Eur J Ophthalmol. 2005 Jan-Feb;15(1):96-101. doi: 10.1177/112067210501500115. PMID 15751246
- [Background] Ozkiris A, Evereklioglu C, Erkilic K, Dogan H. Intravitreal triamcinolone acetonide for treatment of persistent macular oedema in branch retinal vein occlusion. Eye (Lond). 2006 Jan;20(1):13-7. doi: 10.1038/sj.eye.6701803. PMID 15723039
- [Background] Yamamoto S, Saito W, Yagi F, Takeuchi S, Sato E, Mizunoya S. Vitrectomy with or without arteriovenous adventitial sheathotomy for macular edema associated with branch retinal vein occlusion. Am J Ophthalmol. 2004 Dec;138(6):907-14. doi: 10.1016/j.ajo.2004.06.061. PMID 15629280
- [Background] Garcia-Arumi J, Martinez-Castillo V, Boixadera A, Blasco H, Corcostegui B. Management of macular edema in branch retinal vein occlusion with sheathotomy and recombinant tissue plasminogen activator. Retina. 2004 Aug;24(4):530-40. doi: 10.1097/00006982-200408000-00005. PMID 15300073